CLINICAL TRIAL: NCT05894460
Title: Constrained Balloon Combined With Drug-coated Balloon Angioplasty for Femoropopliteal Lesion: a Single-centre, Prospective Observational Study
Brief Title: Constrained Balloon Combined With Drug-coated Balloon Angioplasty for Femoropopliteal Lesion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: Chocolate-FP
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Femoral artery; Popliteal artery; Peripheral artery disease; Chocolate percutaneous transluminal angioplasty balloon; Drug-coated balloon
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Chocolate balloon
  Interventions: Device: Chocolate balloon
- Conventional ballon
  Interventions: Device: Chocolate balloon

INTERVENTIONS:
Device: Chocolate balloon — Vascular preparation with chocolate balloons prior to drug-coated balloon angioplasty

SUMMARY:
This study will assess the safety and efficacy of Chocolate balloons as a combination with drug-coated balloons in the treatment of popliteal artery lesions in lower limb atherosclerotic occlusive disease and will compare them with conventional balloons.

ELIGIBILITY:
Inclusion Criteria:

* Rutherford classification of 2-6 in patients with femoropopliteal atherosclerotic occlusive disease;
* primary cases with no previous surgical treatment of the target lesion;
* presence of at least one vessel with patency in the distal outflow tract;
* survival >1 year.

Exclusion Criteria:

* planned stenting;
* presence of flow-limiting dissection prior to application of Chocolate balloon and conventional balloon dilation of the target lesion;
* combination of severe organ dysfunction of the heart, lungs and brain that cannot tolerate the procedure;
* allergy to contrast agents, anaesthetic drugs, anticoagulants and anti-platelet drugs;
* ineffective recanalization attempts;
* lesions within or adjacent to the aneurysm, or the presence of a popliteal aneurysm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with femoropopliteal atherosclerotic occlusive disease
Sampling Method: Probability Sample
Enrollment: 254 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 12 months
  No occlusion or restenosis (>50%) of the target vessel in the treated segment during follow-up and no further intervention is required.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, None Selected, China

IPD SHARING:
Plan to Share IPD: Undecided